CLINICAL TRIAL: NCT00739908
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel-Group, Assessment of the Efficacy, Safety and Tolerability of CX157 (TriRima) 60mg Three Times a Day (TID) in Subjects With Major Depressive Disorder
Brief Title: A Study of CX157 (TriRima) for the Treatment of Depression
Acronym: CX157-200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CeNeRx BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX157-200
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — CX157; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CX157 (TriRima) (Experimental)
  Interventions: Drug: CX157 (TriRima)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CX157 (TriRima) — Six capsules administered three times a day for six weeks.
  Arms: CX157 (TriRima)
Drug: Placebo — Six capsules administered three times a day for six weeks.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy of CX157 60 mg administered three times a day (180 mg daily dose) as compared to placebo in subjects with Major Depressive Disorder (MDD). Secondary objectives are to evaluate the safety and tolerability and steady state pharmacokinetic profile of CX157 in these subjects.

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled, parallel-group, multi-center study comparing the efficacy, safety and tolerability of CX157 60mg TID and placebo. This study will be conducted at approximately 12 investigative sites in the US.

Subjects with suspected Major Depressive Disorder (MDD) and experiencing a Major Depressive Episode (MDE) who the investigator wishes to consider for enrollment in the study and who provide written informed consent will initially be evaluated by the Inventory of Depressive Symptomatology 30 item -Self Report (IDS-SR30) administered via Interactive Voice Response System (IVRS). Subjects who meet the minimum score of 40 on the IDS-SR30 will proceed with the remaining study related assessments at the Screening visit. Those subjects who meet all inclusion criteria and none of the exclusion criteria will enter a one to two week Screening period to confirm eligibility and to capture Screening data prior to Randomization. At the Randomization visit, all eligibility requirements will be reconfirmed. The subjects who meet all criteria will be randomized to study medication and enter into a six-week treatment period and a subsequent one week Follow-Up period. The total duration of participation for subjects who complete all phases of the study will be approximately 8-9 weeks. During the treatment period, clinic visits will occur at Week 1, Week 2, Week 4, and Week 6. A subsequent clinic visit will occur at the end of the one week Follow-Up period. The clinical site will contact the subjects via telephone at Weeks 3 and 5 to inquire about their wellbeing, query about adverse events and administer the suicidality scale.

Eligible subjects will be randomized (1:1) to receive:

* CX157 60mg three times a day (TID) for a total daily dose of 180 mg, or
* Placebo administered three times a day.

Subjects who discontinue from the study for any reason will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Male or female = 18 years of age and <60 years
* Able to read, understand, converse in English
* Willing to comply with diet restrictions, concomitant medication restrictions, & all study requirements
* Good general health as ascertained by:Medical history, Physical exam, Supine & standing vital signs, Clinical lab evaluations, 12-lead Electrocardiogram (ECG)
* Diagnosis of MDD;
* A total score =>40 on the IDS-SR30 assessed via IVRS at Screening and Randomization

Exclusion Criteria:

* Subject's current MDD episode is >2 years
* History of Substance Use Disorder at Screening or 12 months prior (except for nicotine)
* Current diagnosis of Obsessive-Compulsive Disorder;

  * Panic Disorder or Post-Traumatic Stress Disorder;
  * Anorexia nervosa, Bulimia nervosa, or eating disorder not otherwise specified;
  * Any Axis I Disorder clinically predominant to their MDD (within 6 mo);
  * Presence of psychotic features with current depressive episode;
  * Antisocial or Borderline Personality Disorder
* At risk for suicide
* Lack of response to >2 trials of adequate dose & duration of antidepressants of different mechanistic classes
* Electroconvulsive therapy within 1 year of Screening
* Subject has taken any psychoactive drug within 2 weeks of Randomization
* History of cardiac abnormalities including abnormal vital sign measurements
* Clinically significant abnormal ECG at Screening
* History within past 2 years of: Significant head trauma;

  * Surgical procedure involving brain or meninges; Encephalitis or meningitis;
  * Degenerative CNS disorder (Alzheimer's or Parkinson's);
  * Epilepsy;
  * Mental retardation
* Clinically significant Liver Function Test (LFT) and other lab abnormalities
* A history of hypothyroidism and treatment with a stable dosage of thyroid replacement medication for <6 months prior to Screening
* A history of hyperthyroidism treated (medically or surgically) <6 months prior to Screening
* Participation in a clinical investigation of a psychotropic drug within 90 days prior to Screening OR used any other investigational drug within 60 days prior to Screening
* Presence of any medical history which includes:

  * Hypersensitivity to CX157 or excipients, other MAO inhibitors, or other phenylethylamines;
  * Diabetes mellitus Type I, uncontrolled Type II, or controlled Type II managed with insulin; Malignancy/chemotherapy within 2 years prior to Screening;
  * Malignancy >2 yrs may not preclude participation if the malignancy was local and without metastasis or recurrence and, if treated with chemotherapy, had no nervous system complications (e.g basal cell carcinoma);
  * Pheochromocytoma
* Positive urine test for drugs of abuse (blood for alcohol)
* Female subject who is pregnant or lactating
* Poor likelihood of subject's cooperation or compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burch, MD, Study Director — CeNeRx BioPharma Inc.
Locations (14):
- United States (14):
  - Birmingham Research Group, Birmingham, Alabama
  - Southwestern Research, Inc., Beverly Hills, California
  - The George Washington University, Washington D.C., District of Columbia
  - Irving S. Kolin, M.D., Winter Park, Florida
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - Capital Clinical Research Associates, Rockville, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - CRI Worldwide, LLC, Clementon, New Jersey
  - Fieve Clinical Services, New York, New York
  - Richard H. Weisler, M.D., P.A., Raleigh, North Carolina
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Summit Research Network (Seattle), LLC, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin

REFERENCES:
- [Derived] Targum SD. Early symptomatic improvement affects treatment outcome in a study of major depressive disorder. J Psychiatr Res. 2017 Dec;95:276-281. doi: 10.1016/j.jpsychires.2017.09.009. Epub 2017 Sep 8. PMID 28926793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 out-patient medical centers in the United States (US) from 16 September 2008 (date of first subject randomized) to 09 July 2009 (last subject's last visit).
Pre-assignment Details: A total of 587 subjects were screened. Three hundred and two (302) subjects failed to meet study entry criteria, and thus were screen failures. The top three reasons for screen failure were: IDS-SR30 total score cut-off for randomization not met (204 pts); presence of cardiovascular abnormality (18 pts) and Laboratory Abnormalities (14 pts).
Groups:
- Oral CX157 60 mg TID (Total Daily Dose of 180 mg): CX157 is an investigational compound. The mechanism of action of this compound is Reversible Monoamine oxidase inhibition (MAOI)
- Oral Placebo TID: Placebo does not have any active medication and is the same as a Sugar Pill.
Period: Overall Study
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Started | 142 | 143
Completed | 117 | 118
Not Completed | 25 | 25
Not completed — Adverse Event | 5 | 6
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 14 | 9
Not completed — Non-Compliance With Study Procedures | 2 | 3
Not completed — Non-Compliance With Study Medication | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Relocation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID | Total
Number analyzed (Participants) | 142 | 143 | 285
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 5 | 5
  Between 18 and 65 years | 142 | 138 | 280
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.14) | 38.5 (11.16) | 38.8 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 81 | 161
  Male | 62 | 62 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 32 | 62
  White | 102 | 105 | 207
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 142 | 143 | 285

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization in Montgomery and Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item checklist designed to measure the overall severity of depressive symptoms in patients with MDD [Montgomery, 1979]. Items are rated on a scale of 0-6, with scores ranging from 0 to 60 with 0 being symptom free and 60 being the most severe depression. MADRS was assessed at randomization and Weeks 1, 2, 4 and 6 of the study.
Time Frame: Randomization and study end (Week 6).
Population: mITT population consisted of all patients with at least one post randomzation MADRS score. The primary efficacy variable was the change-from-randomization to each available post-randomization measurement of the MADRS total score, used as the response variable in a mixed model repeated measures (MMRM) analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Oral CX157 60 mg TID (Total Daily Dose of 180 mg): CX157 is an investigational Reversible Monoamine Oxidase Inhibitor (MAOI)
- Oral Placebo TID: No active medication, the same as a Sugar Pill
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
units on a scale | -12.5 [-14.4 to -10.5] | -12.3 [-14.2 to -10.3]

2. Secondary Outcome: Montgomery and Asberg Depression Rating Scale (MADRS) Response Rate
Description: MADRS is a 10-item checklist designed to measure the overall severity of depressive symptoms in patients with MDD [Montgomery, 1979]. Items are rated on a scale of 0-6, with scores ranging from 0 to 60 with 0 being symptom free and 60 being the most severe depression. Percentage of participants who achieved a reduction in total MADRS score of at least 50% or more as compared to baseline. MADRS was assessed at randomization and Weeks 1, 2, 4, and 6 of the study. MADRS Responder rate at Week 6 or the last available post treatment result (LOCF) is reported here.
Time Frame: Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomization MADRS score.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
percentage of participants | 31.7 [24.0 to 40.1] | 34.3 [26.5 to 42.7]

3. Secondary Outcome: Montgomery and Asberg Depression Rating Scale (MADRS) Remitter Rate
Description: Percentage of participants with total MADRS score of 11 or less. MADRS was assessed at randomization and Weeks 1, 2, 4, and 6 of the study. MADRS Remitter rate at Week 6 or the last available post treatment result (LOCF)is reported here.
Time Frame: Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomzation MADRS score.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
Percentage of Participants | 19.4 [13.2 to 27] | 23.1 [16.4 to 30.9]

4. Secondary Outcome: The Hospital Anxiety and Depression Scale (HADS)
Description: HADS is a subject-rated questionnaire designed to detect states of anxiety and depression. The HADS consists of 14 questions relating to anxiety or depression, each with a choice of four responses [Zigmond, 1983]. These responses are numerically scored 0-3, with 0 representing the least severe response and 3 representing the most severe response. The highest possible total score is 42. HADS was assessed at randomization and Weeks 1, 2, 4, and 6 of the study. Change from randomization in the HADS total score at Week 6 or the last available post treatment result (LOCF) is reported here.
Time Frame: Randomization and Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomzation MADRS score.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
units on a scale | -8.7 [-10.1 to -7.2] | -8.9 [-10.3 to -7.5]

5. Secondary Outcome: Inventory of Depressive Symptomatology 30 Item -Self Report (IDS -SR 30 Items)
Description: IDSR-SR 30 measures the severity of depressive symptoms by subjects. This scale has 30 items. The minimum score is 0 and the maximum possible IDS-30 score is 90 (the highest severity). IDS-SR30 was administered at screening, randomization and Weeks 1, 2, 4, and 6. Change from randomization in the IDS-SR30 total score at Week 6 or the last available post treatment result (LOCF) is reported here.
Time Frame: Randomization and Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomzation MADRS score.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
units on a scale | -22.58 [-26.34 to -18.82] | -23.39 [-26.99 to -19.79]

6. Secondary Outcome: Clinical Global Impression - Improvement of Illness (CGI-I)
Description: The Clinical Global Impression - Improvement of Illness (CGI-I) was rated on a 7-point scale by the investigator to measure subject's total improvement compared to his/her condition at randomization according to the following scale: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. CGI-I was measured at Weeks 1, 2, 4 and 6. Percentage of participants "very much improved" and "much improved" at Week 6 or the last available post treatment result (LOCF) is reported here.
Time Frame: Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomzation MADRS score.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
Percentage of Participants | 36.7 | 39.9

7. Secondary Outcome: Clinical Global Impression - Severity of Illness (CGI-S)
Description: CGI-S measures the study rater's assessment of the severity of depression illness. CGI-S is rated on a scale of 1-7 as follows: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = among the most extremely ill patients. CGI-S was measured at randomization and Weeks 1, 2, 4 and 6. Percentage of subjects reported as normal, not at all ill; borderline mentally ill; and mildly ill is reported here at Week 6 or the last available post treatment result (LOCF).
Time Frame: Week 6 or the last available post treatment result (LOCF)
Population: mITT population consisted of all patients with at least one post randomzation MADRS score.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Number analyzed (Participants) | 139 | 143
Percentage of Participants | 36.7 | 39.9

ADVERSE EVENTS:
Time Frame: 16 September 2008 (date of first subject randomized) to 09 July 2009 (last subject's last visit)
Arm/Group | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) | Oral Placebo TID
Serious Adverse Events (participants affected / at risk) | 3/142 | 3/143
Other Adverse Events (participants affected / at risk) | 39/142 | 27/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) (N=142) | Oral Placebo TID (N=143)
Urinary Tract Infection (UTI) (Infections and infestations) | 1 (1) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral CX157 60 mg TID (Total Daily Dose of 180 mg) (N=142) | Oral Placebo TID (N=143)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 6 (6)
Upper Respiratory Tract Infection (URTI) (Infections and infestations) | 8 (8) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8) | 5 (5)

LIMITATIONS AND CAVEATS:
Subjects were asked to take 6 capsules 3 times a day for 6 weeks. Non-adherence with the study medication was high based on the population PK data. This likely contributed to the results in CX157 treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators were informed that the first publication or disclosure of study results shall be a complete, joint multicenter publication or disclosure coordinated by CeNeRx. Thereafter, any secondary publications will reference the original publication(s).